CLINICAL TRIAL: NCT00005155
Title: Physiological and Psychosocial Correlates of Type A Behavior
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1027; R01HL028094 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To test the physiological and psychosocial correlates of Type A behavior.

DETAILED DESCRIPTION:
BACKGROUND:

The Type A behavior pattern as described by Friedman and Rosenman is characterized by extremes of competitiveness, easily aroused hostility, a sense of urgency and aggression. In 1981 the Review Panel of Coronary Prone Behavior and Coronary Heart Disease concluded that the Type A behavior pattern was associated with an increased risk for coronary heart disease. Studies have challenged the independent predictive value of the behavior pattern with respect to coronary heart disease. There was a need to develop physiological measurements related to coronary-prone behavior and to reexamine the stability of the psychological assessment. It was hypothesized that Type A behavior or some component such as hostility might be associated with a state of chronic, generalized sympathetic-adrenal arousal. Preliminary research was conducted on interpersonal dynamic correlates of Type A behavior among married couples. Research was needed on whether certain types of marriages, according to the Type A/B classification of the two spouses, are more pathogenic than others. Additional research is also needed on which components of the global Type A pattern were of primary importance as risk factors for coronary disease, and which components were enduring, which were transient, and which were situationally related.

In 1982, a household survey on Type A behavior was initiated. Measures included the Jenkins Activity Survey, the Framingham Type A Questionnaire, hostility scales, and other behavioral tests. Information was also collected on demographic variables, social support, marital satisfaction, life events, social values, and job and family stress. After the household survey was completed, the respondents were contacted by the Type A interviewers and the Structured Interviews conducted. A total of 1,114 Type A interviews were completed yielding 902 primary respondents and 239 spouses.

DESIGN NARRATIVE:

The concurrent relationship of the Structured Interview (SI) global and component Type A behavior measures were tested to levels of chronic and acute sympathetic nervous system activity, as assessed by platelet and plasma catecholamines, heart rate, blood pressure, and pupil size. The correlations among heart rate, pupil size, blood pressure, and the plasma and platelet catecholamine measures were determined as were the relationships with reported global health, chronic disease, and functional disability levels. The five-year predictability was tested of reported global health, chronic disease, and functional disability from measures of global and component Type A behavior.

Tests were made of the differences in the chronic and acute sympathetic-adrenal responses, as assessed by platelet and plasma catecholamines, pupil size, heart rate, and blood pressure, among married couples having different combinations of Structured Interview global and component Type A classifications. The five year marital stability and health of these couples were followed. A comparison was made of one week test-retest reliability with the five year stability of the Structured Interview global and component Type A measures.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1982-02; Study Completion 1989-01 (Actual)

REFERENCES:
- [Background] Harlan WR: Rationale for Intervention on Blood Pressure in Childhood and Adolescence. In: Matarazzo JD, Weiss SM, Herd JA, (Eds), Behavioral Health: A Handbook of Health Enhancement and Disease Prevention. New York: Wiley & Sons, 1984
- [Background] Moss GE, Dielman TE, Campanelli PC, Leech SL, Harlan WR, Harrison RV, Horvath WJ. Demographic correlates of SI assessments of type A behavior. Psychosom Med. 1986 Nov-Dec;48(8):564-74. doi: 10.1097/00006842-198611000-00003. PMID 3809368
- [Background] Dielman TE, Butchart AT, Moss GE, Harrison RV, Harlan WR, Horvath WJ. Psychometric properties of component and global measures of structured interview assessed type A behavior in a population sample. Psychosom Med. 1987 Sep-Oct;49(5):458-69. doi: 10.1097/00006842-198709000-00003. PMID 3671635
- [Background] Cwikel JM, Dielman TE, Kirscht JP, Israel BA. Mechanisms of psychosocial effects on health: the role of social integration, coping style and health behavior. Health Educ Q. 1988 Summer;15(2):151-73. doi: 10.1177/109019818801500202. PMID 3378901